CLINICAL TRIAL: NCT01397669
Title: Characteristics of Immunity in Gut Mucosa, Spinal Fluid, Lymph Node and Blood of HIV Negative Thais and Thais with HIV Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEARCH Research Foundation (Other)
Collaborators: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government); Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Principal Investigator, Nittaya Phanuphak, Exceutive director of IHRI, Institute of HIV Research and Innovation Foundation, Thailand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WRAIR#1751 /RV304/ SEARCH013
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: HIV-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Spinal Puncture; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV infection and non HIV infection (Other)
  Interventions: Procedure: Colon biopsy, lymph node biopsy, lumbar puncture, Leukapheresis, Brain MRI/MRS/DTI

INTERVENTIONS:
Procedure: Colon biopsy, lymph node biopsy, lumbar puncture, Leukapheresis, Brain MRI/MRS/DTI — Eligible subjects will undergo a flexible sigmoidoscopy/biopsy and Brain MRI/MRS/DTI at Chulalongkorn University Hospital.
  Lumbar puncture, lymph node biopsy, and leukapheresis will be done at TRCARC or IHRI.

SUMMARY:
To compare the immunophenotyping and immunochemistry in the gut mucosa of HIV negative and non-acute HIV-infected adults

1. To compare the immunophenotyping of the gut mucosa to that of the peripheral blood in HIV negative and in non-acute HIV-infected subjects
2. To compare the immunophenotyping of the peripheral blood in HIV negative and non-acute HIV-infected adults to the findings from acutely HIV-infected subjects in the WRAIR#1494/RV254/ SEARCH 010 study
3. To compare immunologic markers in the genital compartment compared to the peripheral blood in HIV negative and non-acute HIV-infected adults to the findings from acutely HIV-infected subjects in the WRAIR#1494/RV254/ SEARCH 010 study
4. Archive samples for immunologic and virologic testing

DETAILED DESCRIPTION:
This study will provide control samples for immunologic and virologic investigations from HIV negative and non-acute HIV-infected subjects to compare to subjects with acute HIV infection in WRAIR#1494/RV254/SEARCH 010 study. These control samples will allow for correct scientific interpretation of the immunologic changes seen in acute HIV infection in the peripheral blood, gut and genital compartments.

Subjects will be recruited at the Thai Red Cross Anonymous Clinic (TRCAC) and Chulalongkorn University Hospital. Eligible subjects will undergo a one-time flexible sigmoidoscopy and biopsy at Chulalongkorn University Hospital. They will have a total of approximately 60 ml of blood draw for immunophenotyping and storage. Genital secretion will be collected in subjects who agree to this optional procedure.

It will take approximately 12 months to complete the study. Each subject will have two visits: the screening visit and the enrollment visit (within 15 days of screening visit). Subjects may also be co-enrolled in other study protocols provided blood volumes are within acceptable limits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years old
2. HIV negative subjects must have negative results by 4th generation EIA and NAT (Aptima)
3. HIV positive subjects must have a positive 4th generation EIA and a positive less sensitive EIA.
4. Understand the study and sign informed consent form. Persons who cannot read will have the consent form read to them by a study staff and they can give informed consent by using thumb print.

Exclusion Criteria:

1. Have gastrointestinal disorders or gastrointestinal symptoms that require endoscopy for diagnostic purposes or have systemic disorders, which include but may not be limited to autoimmune diseases such as rheumatoid arthritis, systemic lupus erythematosus or psoriasis, that in the judgment of investigators could cause colon mucosa to be abnormal on biopsy
2. Active AIDS-defining opportunistic infection (OI) within 30 days prior to entry for HIV-positive subjects. Subjects must be off all acute treatments for OI for at least 14 days prior to entry. Subjects on maintenance or prophylactic therapy for AIDS-related OIs will be eligible.
3. Have platelet count < 150,000 count/ml or PT, PT/PTT > the upper limit of normal (ULN) or INR > 1.1
4. Have self-reported bleeding disorder
5. Untreated syphilis infection
6. Abnormal screening neurological examination suggestive of central neurological findings if planning to participate in the lumbar puncture
7. Positive urine pregnancy test
8. Persons who have a history of a medical or psychiatric disorder by investigator's interview and physical examination according to standard practices, that in the judgment of the investigator(s), would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 214 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Number of HIV and non-HIV related clinical events | It will take approximately 24 months to complete the study.

SECONDARY OUTCOMES:
the immunophenotyping of the gut mucosa | Approximately 24 months to complete the study.
the immunophenotyping of the peripheral blood | approximately 24 months to complete the study
immunologic markers in the genital compartment | approximately 24 months to complete the study
the immunophenotyping of the CSF | approximately 24 months to complete the study
immunologic markers in the lymph node | approximately 24 months to complete the study

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of HIV Research and Innovation (IHRI), Bangkok, Bangkok, Thailand